CLINICAL TRIAL: NCT01576523
Title: An Open-label, Cross-over, Dose-ranging Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of the Subcutaneous Administration of a Human Plasma-derived C1-esterase Inhibitor in Subjects With Hereditary Angioedema
Brief Title: A Study to Evaluate the Clinical Pharmacology and Safety of C1-esterase Inhibitor Administered by the Subcutaneous Route
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CSL830_2001; 2011-005013-36 (EudraCT Number)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hereditary Angioedema Types I and II
MeSH Terms: conditions — Hereditary Angioedema Types I and II

ARMS (6):
- Low, then medium, C1-esterase inhibitor dose (Experimental)
  Interventions: Biological: C1-esterase inhibitor - single intravenous dose; Biological: C1-esterase inhibitor - subcutaneous low dose; Biological: C1-esterase inhibitor - subcutaneous medium dose
- Medium, then low, C1-esterase inhibitor dose (Experimental)
  Interventions: Biological: C1-esterase inhibitor - single intravenous dose; Biological: C1-esterase inhibitor - subcutaneous low dose; Biological: C1-esterase inhibitor - subcutaneous medium dose
- Medium, then high, C1-esterase inhibitor dose (Experimental)
  Interventions: Biological: C1-esterase inhibitor - single intravenous dose; Biological: C1-esterase inhibitor - subcutaneous medium dose; Biological: C1-esterase inhibitor - subcutaneous high dose
- Low, then high, C1-esterase inhibitor dose (Experimental)
  Interventions: Biological: C1-esterase inhibitor - single intravenous dose; Biological: C1-esterase inhibitor - subcutaneous low dose; Biological: C1-esterase inhibitor - subcutaneous high dose
- High, then low, C1-esterase inhibitor dose (Experimental)
  Interventions: Biological: C1-esterase inhibitor - single intravenous dose; Biological: C1-esterase inhibitor - subcutaneous low dose; Biological: C1-esterase inhibitor - subcutaneous high dose
- High, then medium, C1-esterase inhibitor dose (Experimental)
  Interventions: Biological: C1-esterase inhibitor - single intravenous dose; Biological: C1-esterase inhibitor - subcutaneous medium dose; Biological: C1-esterase inhibitor - subcutaneous high dose

INTERVENTIONS:
Biological: C1-esterase inhibitor - single intravenous dose — A single intravenous dose of C1-esterase inhibitor (Berinert) at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor.
Biological: C1-esterase inhibitor - subcutaneous low dose — A low dose of C1-esterase inhibitor will be administered subcutaneously twice a week for four weeks.
  Arms: High, then low, C1-esterase inhibitor dose; Low, then high, C1-esterase inhibitor dose; Low, then medium, C1-esterase inhibitor dose; Medium, then low, C1-esterase inhibitor dose
Biological: C1-esterase inhibitor - subcutaneous medium dose — A medium dose of C1-esterase inhibitor will be administered subcutaneously twice a week for four weeks.
  Arms: High, then medium, C1-esterase inhibitor dose; Low, then medium, C1-esterase inhibitor dose; Medium, then high, C1-esterase inhibitor dose; Medium, then low, C1-esterase inhibitor dose
Biological: C1-esterase inhibitor - subcutaneous high dose — A high dose of C1-esterase inhibitor will administered subcutaneously twice a week for four weeks.
  Arms: High, then low, C1-esterase inhibitor dose; High, then medium, C1-esterase inhibitor dose; Low, then high, C1-esterase inhibitor dose; Medium, then high, C1-esterase inhibitor dose

SUMMARY:
The aim of the study is to assess what happens to C1-esterase inhibitor that is administered under the skin of subjects with hereditary angioedema. Three different dosing regimens of C1-esterase inhibitor will be assessed. Each subject will be assigned to receive 2 of the 3 dosing regimens, each for 4 weeks. The activity and concentration of C1-esterase inhibitor in the blood will be measured during each 4-week period. The study will also examine how well C1-esterase inhibitor administered under the skin is tolerated by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older.
* Laboratory-confirmed hereditary angioedema type I or II.
* Less than two hereditary angioedema attacks per month in the last three months.
* Body weight of 50.0 kg to 110.0 kg.

Exclusion Criteria:

* Receiving prophylactic C1-esterase inhibitor therapy.
* Received C1-esterase inhibitor, ecallantide, icatibant or any blood products for the prevention or treatment of hereditary angioedema within 7 days before the screening visit.
* Intends to use recombinant C1-esterase inhibitor or fresh frozen plasma for the acute treatment of hereditary angioedema during the study.
* Received androgen therapy (e.g., danazol, oxandrolone, stanozolol, testosterone) within 30 days before the screening visit.
* Female subjects who started taking or changed dose of any hormonal contraceptive regimen or hormone replacement therapy (i.e., estrogen/progesterone-containing products) within 3 months prior to the screening visit.
* Known or suspected hypersensitivity to the study product, or to any excipients of the study product.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Program Director, Study Director — CSL Behring
Locations (8):
- United States (5):
  - Study Site, Atlanta, Georgia
  - Study Site, Chevy Chase, Maryland
  - Study Site, Cincinnati, Ohio
  - Study Site, Toledo, Ohio
  - Study Site, Hershey, Pennsylvania
- Germany (3):
  - Study Site, Berlin
  - Study Site, Frankfurt
  - Study Site, Mainz

REFERENCES:
- [Result] Zuraw BL, Cicardi M, Longhurst HJ, Bernstein JA, Li HH, Magerl M, Martinez-Saguer I, Rehman SM, Staubach P, Feuersenger H, Parasrampuria R, Sidhu J, Edelman J, Craig T. Phase II study results of a replacement therapy for hereditary angioedema with subcutaneous C1-inhibitor concentrate. Allergy. 2015 Oct;70(10):1319-28. doi: 10.1111/all.12658. Epub 2015 Aug 11. PMID 26016741

RESULTS

PARTICIPANT FLOW:
Groups:
- Low, Then Medium, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1-esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830).
  C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1-esterase inhibitor (1500 IU) will be administered subcutaneously twice a week for four weeks, then
  C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks.
- Medium, Then Low, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1-esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830).
  C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks, then
  C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1-esterase inhibitor (1500 IU) will be administered subcutaneously twice a week for four weeks.
- Medium, Then High, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1-esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830).
  C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks, then
  C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will administered subcutaneously twice a week for four weeks.
- Low, Then High, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1-esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830).
  C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1-esterase inhibitor (1500 IU) will be administered subcutaneously twice a week for four weeks, then
  C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will administered subcutaneously twice a week for four weeks.
- High, Then Low, CSL830 Dose: C1-esterase inhibitor - single intravenous dose:(Berinert): A single intravenous dose of C1-esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830).
  C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will be administered subcutaneously twice a week for four weeks, then
  C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1-esterase inhibitor (1500 IU) will administered subcutaneously twice a week for four weeks.
- High, Then Medium, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1-esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830).
  C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will be administered subcutaneously twice a week for four weeks, then
  C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks.
Period: Dosing Period 1
Arm/Group | Low, Then Medium, CSL830 Dose | Medium, Then Low, CSL830 Dose | Medium, Then High, CSL830 Dose | Low, Then High, CSL830 Dose | High, Then Low, CSL830 Dose | High, Then Medium, CSL830 Dose
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dosing Period 2
Arm/Group | Low, Then Medium, CSL830 Dose | Medium, Then Low, CSL830 Dose | Medium, Then High, CSL830 Dose | Low, Then High, CSL830 Dose | High, Then Low, CSL830 Dose | High, Then Medium, CSL830 Dose
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low, Then Medium, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1- esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830). C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1- esterase inhibitor (1500 IU) will be administered subcutaneously twice a week for four weeks, then C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks.
- Medium, Then Low, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1- esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830). C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks, then C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1- esterase inhibitor (1500 IU) will be administered subcutaneously twice a week for four weeks.
- Medium, Then High, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1- esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830). C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks, then C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will administered subcutaneously twice a week for four weeks.
- Low, Then High, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1- esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830). C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1- esterase inhibitor (1500 IU) will be administered subcutaneously twice a week for four weeks, then C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will administered subcutaneously twice a week for four weeks.
- High, Then Low, CSL830 Dose: C1-esterase inhibitor - single intravenous dose:(Berinert): A single intravenous dose of C1- esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830). C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will be administered subcutaneously twice a week for four weeks, then C1-esterase inhibitor - subcutaneous low dose (CSL830): A low dose of C1- esterase inhibitor (1500 IU) will administered subcutaneously twice a week for four weeks.
- High, Then Medium, CSL830 Dose: C1-esterase inhibitor - single intravenous dose(Berinert): A single intravenous dose of C1- esterase inhibitor at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor (CSL830). C1-esterase inhibitor - subcutaneous high dose (CSL830): A high dose of C1-esterase inhibitor (6000 IU) will be administered subcutaneously twice a week for four weeks, then C1-esterase inhibitor - subcutaneous medium dose (CSL830): A medium dose of C1-esterase inhibitor (3000 IU) will be administered subcutaneously twice a week for four weeks.
- Total: Total of all reporting groups
Arm/Group | Low, Then Medium, CSL830 Dose | Medium, Then Low, CSL830 Dose | Medium, Then High, CSL830 Dose | Low, Then High, CSL830 Dose | High, Then Low, CSL830 Dose | High, Then Medium, CSL830 Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 3 | 3 | 3 | 17
  >=65 years | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 2 | 2 | 11
  Male | 1 | 1 | 2 | 1 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Modeled C1-esterase Inhibitor Functional Activity Trough Level
Description: Mean trough C1-esterase inhibitor functional activity of the low, medium and high subcutaneous dose regimens, based on modeling and simulation
Time Frame: at the fourth week of each dosing regimen
Population: Complete Analysis Set (CAS) - Subjects received at least 1 dose (complete or incomplete) of the dosing regimen of CSL830 and provided at least 1 C1-INH functional activity measurement during the dosing regimen (prior to the use of any prohibited concomitant therapy or prohibited change in dosage of a concomitant therapy)
Measure: Mean (Standard Deviation); unit: percent functional activity
Groups:
- CSL830 (Low Dose): A low dose of C1-esterase inhibitor (1500 IU) administered subcutaneously twice a week for four weeks
- CSL830 (Medium Dose): A medium dose of C1-esterase inhibitor (3000 IU) administered subcutaneously twice a week for four weeks
- CSL830 (High Dose): A high dose of C1-esterase inhibitor (6000 IU) administered subcutaneously twice a week for four weeks
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 12 | 12
percent functional activity | 30.3 (9.07) | 45.9 (14.35) | 80.6 (23.47)

2. Secondary Outcome: As-observed C1-esterase Inhibitor Functional Activity Trough Level
Description: Mean trough C1-esterase inhibitor functional activity of the low, medium and high subcutaneous dose regimens
Time Frame: during the last week of 4-week dose regimen
Population: As-observed analysis set - subset of the full analysis set (FAS). FAS consisted of all enrolled subjects (all subjects who gave informed consent).
Measure: Mean (Standard Deviation); unit: percent functional activity
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 11 | 12
percent functional activity | 31.7 (9.97) | 44.3 (17.73) | 80.5 (24.92)

3. Secondary Outcome: C1-esterase Inhibitor Concentration Trough Level
Description: Mean trough C1-esterase inhibitor concentration of the low, medium and high subcutaneous dose regimens
Time Frame: during the last week of 4-week dose regimen
Population: As-observed analysis set
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 11 | 12
mg/mL | 0.06 (0.024) | 0.15 (0.130) | 0.23 (0.158)

4. Secondary Outcome: C4 Concentration Trough Level
Description: Mean trough C4 concentration of the low, medium and high subcutaneous dose regimens
Time Frame: during the last week of 4-week dose regimen
Population: As-observed analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 11 | 12
mg/dL | 11.1 (4.45) | 14.1 (5.28) | 18.4 (6.55)

5. Secondary Outcome: Change From Baseline in C1-esterase Inhibitor Functional Activity
Description: Mean change from baseline of C1-esterase inhibitor functional activity of the low, medium and high subcutaneous dose regimens
Time Frame: Baseline and during the last week of 4-week dose regimen
Population: As-observed analysis set
Measure: Mean (Standard Deviation); unit: percent functional activity
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 11 | 12
percent functional activity | 16.4 (7.41) | 33.2 (11.32) | 63.3 (21.33)

6. Secondary Outcome: Change From Baseline in C1-esterase Inhibitor Concentration
Description: Mean change from baseline of C1-esterase inhibitor concentration of the low, medium and high subcutaneous dose regimens
Time Frame: Baseline and during the last week of 4-week dose regimen
Population: As-observed analysis set
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 11 | 12
mg/mL | 0.02 (0.018) | 0.05 (0.029) | 0.14 (0.047)

7. Secondary Outcome: Change From Baseline in C4 Concentration
Description: Mean change from baseline of C4 concentration of the low, medium and high subcutaneous dose regimens
Time Frame: Baseline and during the last week of 4-week dose regimen
Population: As-observed analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
Number analyzed (Participants) | 12 | 11 | 12
mg/dL | 4.3 (3.00) | 5.6 (11.90) | 9.1 (10.89)

ADVERSE EVENTS:
Time Frame: Up to 14 weeks per subject
Description: The safety set consisted of all enrolled subjects who received at least 1 dose (complete or incomplete) of study drug (Berinert or CSL830). Subjects were included in the safety set for a dosing regimen only if they received at least 1 dose of that dosing regimen (e.g., a subject who discontinued prior to taking the dosing period 2 dosing regimen was not included in the safety set for that dosing regimen).
Groups:
- Berinert: C1-esterase inhibitor - single intravenous dose: A single intravenous dose of C1-esterase inhibitor (Berinert) at 20 units per kg body weight will be administered to all subjects prior to receiving the first dose of subcutaneous C1-esterase inhibitor.
Arm/Group | Berinert | CSL830 (Low Dose) | CSL830 (Medium Dose) | CSL830 (High Dose)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/12 | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 4/18 | 10/12 | 8/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berinert (N=18) | CSL830 (Low Dose) (N=12) | CSL830 (Medium Dose) (N=12) | CSL830 (High Dose) (N=12)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berinert (N=18) | CSL830 (Low Dose) (N=12) | CSL830 (Medium Dose) (N=12) | CSL830 (High Dose) (N=12)
Injection site erythema (General disorders) | 0 (0) | 2 (5) | 2 (3) | 5 (19)
Injection site pain (General disorders) | 0 (0) | 5 (13) | 0 (0) | 2 (12)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 (2) | 2 (9) | 2 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ovarian Cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine spasm (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.